CLINICAL TRIAL: NCT01287338
Title: A Randomized, Double-Masked, Placebo-Controlled, Proof of Concept Study to Evaluate the Short-term Safety and Efficacy of the QLT Proprietary Olopatadine Punctal Plug Delivery System in Subjects With Seasonal Allergic Conjunctivitis to Ragweed in an Environmental Exposure Chamber Model.
Brief Title: A Study to Evaluate the Safety and Efficacy of the QLT Proprietary Olopatadine-PPDS in Subjects With Seasonal Allergic Conjunctivitis to Ragweed in an Environmental Exposure Chamber Model.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of definitive clinical results.
Sponsor: Mati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PP0 AC 01; 141741 (Other: Health Canada: Therapeutic Products Directorate)
Record Dates: First submitted 2011-01-27; First posted 2011-02-01 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Seasonal Allergic Conjunctivitis to Ragweed
MeSH Terms: interventions — Olopatadine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lower Puncta Delivery (Experimental)
  Interventions: Drug: Olopatadine
- Double Puncta Delivery (Experimental)
  Interventions: Drug: Olopatadine

INTERVENTIONS:
Drug: Olopatadine — low dose
  Arms: Lower Puncta Delivery
Drug: Olopatadine — high dose
  Arms: Double Puncta Delivery

SUMMARY:
The purpose of this study is to test if olopatadine punctal plugs can reduce the symptoms (itching) of allergic conjunctivitis to ragweed in an Environmental Exposure Chamber model.

ELIGIBILITY:
Inclusion Criteria:

* History of allergic conjunctivitis to ragweed for at least one year
* Positive skin prick test to ragweed pollen within 12 months prior to visit 1
* BCVA of at leat 20/400

Exclusion Criteria:

* Structural lid abnormalities (ectropion, entropion)
* Active lid disease ( ie moderate or severe blepharitis, meibomianitis) that requires medical treatment
* Presence of follicular conjunctivitis, anterior uveitis or preauricular lymphadenopathy
* History of ophthalmic abnormality, including a history of dry eye
* Perennial allergic rhinoconjunctivitis having significant allergy to animal dander that cannot be avoided during the study period
* History of chronic bacterial or viral ocular infection, such as herpes keratitis, and/or presence of active bacterial or viral ocular infection
* presence of mucous discharge, excess lacrimation or burning as a symptoms of ocular disease
* Currently on any chronic ocular topical medications
* Use of topical or systemic ocular medications during the study period
* History of complications, adverse events, trauma or disease in the nasolacrimal area
* History of symptomatic epiphoria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2010-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Safety of olopatadine-PPDS in subjects with seasonal allergic conjunctivitis to ragweed | 4 Days
Change from baseline in subject-rated ocular itching scores in treated vs placebo control arms in subjects with seasonal allergic conjunctivitis to ragweed | 4 days

SECONDARY OUTCOMES:
Change from baseline and observed values in subject rated ocular itching scores compared between lower puncta delivery and double puncta delivery arms | 4

CONTACTS AND LOCATIONS:
Overall Officials: Dipak Panigrahi, MD, Study Director — QLT Inc.; Deepen Patel, MD, Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Cetero Research, Toronto, Ontario, Canada